CLINICAL TRIAL: NCT00480740
Title: The Pharmacology of Dexmedetomidine in Children With Congenital Heart Disease
Brief Title: The Pharmacology and Hemodynamics of Dexmedetomidine in Children With Congenital Heart Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Julia Finkel, MD, Children's National Research Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB# 3908
Record Dates: First submitted 2007-05-29; First posted 2007-05-31 (Estimated); Results first posted 2015-06-26 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Cardiac Transplant; Patent Ductus Arterious; Atrial Septal Defect; Bidirectional Cavopulmonary Anastomosis
Keywords: Dexmedetomidine; Congenital heart disease; pharmacokinetics; pharmacodynamics; pediatric; Bidirectional cavopulmonary anastomosis; Fontan physiology; Cardiac transplant
MeSH Terms: conditions — Heart Septal Defects, Atrial; Heart Defects, Congenital | interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cardiac Transplant (Experimental): diagnostic cardiac catheterization in children with a transplanted heart
  Interventions: Drug: Dexmedetomidine
- Fontan procedure (Experimental): diagnostic cardiac catheterization in children with a transplanted ventricle
  Interventions: Drug: Dexmedetomidine
- Normal Physiology (Other): diagnostic cardiac catheterization in children with normal cardiac physiology
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine load of 1 microgram/kilogram over 10 minutes, followed by a 1 microgram/kilogram/hour infusion during the time of catheterization
  Other Names: Precedex

SUMMARY:
The purpose of this study is to examine the pharmacokinetics, pharmacodynamics, and pharmacogenomics of dexmedetomidine in the following three pediatric patient populations: patients with bi-directional cavopulmonary anastomosis or a Fontan procedure, patients who have had a cardiac transplant, and patients with otherwise normal physiology who are undergoing closure of a patent ductus arteriosis or atrial septal defect.

DETAILED DESCRIPTION:
While opioid analgesia is currently the mainstream for management of pain in the perioperative setting, it often leads to significant morbidity, including opioid tolerance and hyperalgesia. Looking at ways to decrease the need for opioids with the use of adjunct medications allows for the long-term goal of decreasing physiologic tolerance in children. This is especially relevant in the pediatric congenital heart population.

Dexmedetomidine is in a class of drugs known as alpha-2 agonists and is known to provide analgesia, attenuate opioid tolerance and inhibit the sympathetic stress response. While there are numerous published case studies of dexmedetomidine validating its effectiveness and safety, the pharmacologic and pharmacodynamic profile has not been established.

This study will examine the hemodynamics, pharmacokinetics, and pharmacogenomics of dexmedetomidine in patients with congenital heart disease. The dose-ranging effect of dexmedetomidine will also be investigated. The three groups being studied will be: patients with bi-directional cavopulmonary anastomosis or a Fontan procedure, patients who have had a cardiac transplant, and patients with otherwise normal physiology who are undergoing closure of a patent ductus arteriosis or atrial septal defect.

Comparison: Compare both invasive and noninvasive hemodynamic parameters at baseline sevoflurane and during maintenance dosing on dexmedetomidine. The pharmacokinetics of dexmedetomidine in the pediatric population following escalating loading doses and continuous infusion at timed intervals will be estimated. The efficacy of dexmedetomidine will be estimated by the amount of rescue doses of propofol that are given.

ELIGIBILITY:
Inclusion Criteria:

* age is birth to 18 years
* > or = 6 kg.
* American Society of Anesthesiology (ASA) I, II, or III
* undergone prior cardiac transplant, Fontan or has a patent ductus arterious or atrial septal defect.
* scheduled for cardiac catheterization

Exclusion Criteria:

* subject or family history of malignant hyperthermia
* known hepatic disorder determined by history physical exam or laboratory tests
* pregnant or lactating female
* receiving inotropic agents or has a pacemaker
* weighs less than 6 kg.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 2006-12; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julia C Finkel, MD, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Medical Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Finkel JC, Johnson YJ, Quezado ZM. The use of dexmedetomidine to facilitate acute discontinuation of opioids after cardiac transplantation in children. Crit Care Med. 2005 Sep;33(9):2110-2. doi: 10.1097/01.ccm.0000178183.21883.23. PMID 16148487
- [Background] Finkel JC, Elrefai A. The use of dexmedetomidine to facilitate opioid and benzodiazepine detoxification in an infant. Anesth Analg. 2004 Jun;98(6):1658-1659. doi: 10.1213/01.ANE.0000113547.34160.A5. PMID 15155322

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from cardiology outpatient clinic. The study is anticipating to enroll 104 patients.
Pre-assignment Details: 74 subjects assessed for eligibility, 9 were excluded; 12 did not meet inclusion criteria; 12 refused to enroll; resulting in 41 subjects enrolled
Groups:
- Fontan Physiology: diagnostic cardiac catheterization in children with a transplanted ventricle
Period: Overall Study
Arm/Group | Normal Physiology | Cardiac Transplant | Fontan Physiology
Started | 26 | 9 | 6
Completed | 26 | 9 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Physiology | Cardiac Transplant | Fontan Physiology | Total
Number analyzed (Participants) | 26 | 9 | 6 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.3 (4) | 11 (4.5) | 5.5 (3.3) | 6.9 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 3 | 2 | 22
  Male | 9 | 6 | 4 | 19
Weight (kg) [Mean (Standard Deviation); unit: kg] | 19.1 (14.3) | 35.2 (17.8) | 21.4 (8.7) | 27.3 (13.6)
American Society of Anesthesiology (ASA) physical status classification [Number; unit: participants] — Category 1 means healthy patient Category 2 means mild systemic disease Category 3 means severe systemic disease
  participants
    ASA 1 | 18 | 0 | 0 | 18
    ASA 2 | 8 | 9 | 0 | 17
    ASA 3 | 0 | 0 | 6 | 6
Primary diagnosis [Number; unit: participants]
  ASD | 10 | 0 | 0 | 10
  PDA | 16 | 0 | 0 | 16
  PA with IVS | 0 | 2 | 0 | 2
  HLHS | 0 | 2 | 2 | 4
  Unbalanced AVC | 0 | 1 | 0 | 1
  Cardiomyopathy | 0 | 4 | 0 | 4
  Tricuspid Atresia | 0 | 0 | 2 | 2
  DORV | 0 | 0 | 1 | 1
  Ebstein's anomaly | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Changes in Hemodynamic Variables Recorded During Administration of Sevoflurane + Dexmedetomidine.
Description: Non-inferiority was shown when differences at steady-state (dexmedetomidine + sevoflurane) compared to baseline (sevoflurane alone) and its associated 95% confidence interval fell completely within the range of plus or minus 20%.The 95% confidence interval was normalized by subtracting the baseline values.
  Bispectral Index: monitors electroencephalographic and electromyographic parameters to monitor the depth of anesthesia.
Time Frame: Up to 24 hours following cardiac catheterization
Measure: Mean (95% Confidence Interval); unit: percentage of change from baseline
Arm/Group | Normal Physiology | Cardiac Transplant | Fontan Physiology
Number analyzed (Participants) | 26 | 9 | 6
percentage of change from baseline
  Heart Rate | -0.14 [-0.15 to -0.13] | -0.16 [-0.2 to -0.12] | -0.21 [-0.22 to -0.2]
  Systolic Pressure | 0.15 [0.07 to 0.23] | 0.18 [0.08 to 0.28] | 0.22 [0.16 to 0.28]
  Diastolic Pressure | 0.23 [0.13 to 0.36] | 0.19 [0.13 to 0.25] | 0.09 [-0.11 to 0.29]
  Mean Pressure | 0.23 [0.17 to 0.29] | 0.16 [0.03 to 0.29] | 0.08 [-0.09 to 0.25]
  Bispectral Index | 0.04 [-0.03 to 0.11] | 0.16 [-0.11 to 0.43] | -0.14 [-0.42 to 0.13]
Statistical Analysis 1: Comparison: Normal Physiology vs Cardiac Transplant vs Fontan Physiology; Test type: Non-Inferiority or Equivalence — Noninferiority of dexmedetomindine plus sevoflurane compared with the baseline (sevoflurane alone) for any given variable was reached when the difference (steady-state [dexmedetomidine + sevoflurane]-baseline [sevoflurane0]/baseline [sevoflurane]0 and its associated 95% confidence interval (CI) fell completely withing the range of +/-20% indicated by the gray column; p = 0.05, t-test, 2 sided — The original study design was powered to achieve at least 80% power to detect noninferiority with the two-tailed alpha level set at 0.05 for data with two measurements

ADVERSE EVENTS:
Time Frame: from study start through followup
Groups:
- Normal Physiology: control group
  Dexmedetomidine: Dexmedetomidine load of 1 microgram/kilogram over 10 minutes, followed by a 1 microgram/kilogram/hour infusion during the time of catheterization
Arm/Group | Cardiac Transplant | Fontan Procedure | Normal Physiology
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/6 | 0/26
Other Adverse Events (participants affected / at risk) | 0/9 | 0/6 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No